CLINICAL TRIAL: NCT02808936
Title: The Effect of Remote Ischemic Preconditioning on Major Organ Function in Patients With Coronary Artery Disease Undergoing Orthopedic Surgery - a Randomized Controlled Trial
Brief Title: The Effect of Remote Ischemic Preconditioning on Major Organ Function in Patients With Coronary Artery Disease Undergoing Orthopedic Surgery
Acronym: RIPC-Angina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1604-079-754
Record Dates: First submitted 2016-06-14; First posted 2016-06-22 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Angina Pectoris; Myocardial Infarction
Keywords: remote ischemic conditioning; orthopedic surgery; ischemic heart disease
MeSH Terms: conditions — Angina Pectoris; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC group (Experimental): remote ischemic conditioning group with three cycles of ischemia (5 min) / reperfusion (5 min) of upper or lower limb available with automated RIPC machine using blood pressure cuff
  Interventions: Procedure: Remote ischemic preconditioning
- Control group (Sham Comparator): No remote ischemic conditioning, but blood pressure cuff applied to the upper or lower limb available
  Interventions: Procedure: Sham control

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — three cycles of ischemia (5 min) / reperfusion (5 min) of available upper or lower limb with an automated machine using blood pressure cuff
  Arms: RIPC group
Procedure: Sham control — The patients had the same pneumatic cuff around the upper arm and similar maneuvers were performed, but pressure was not applied to the cuff.
  Arms: Control group

SUMMARY:
The investigators attempt to investigate the organ protective effect of remote ischemic conditioning in patients undergoing non-cardiac surgery with history of ischemic heart disease.

DETAILED DESCRIPTION:
When adult patients with ischemic heart disease undergo non-cardiac surgery, perioperative ischemic complication may occur. These morbidity results in poor clinical outcomes. The incidence of perioperative myocardial ischemic event has been reported to be up to 19.7%. Remote ischemic preconditioning (RIPC) is a concept that a brief ischemic reperfusion of upper or lower extremity can transfer protection to the other vital organs from sustained ischemic reperfusion injury. Although RIPC is extensively studied in high risk cardiovascular surgery, it has not been tested in a non-cardiac surgery patients with a history of ischemic heart disease. Major organ injury including heart, lung and kidney will be evaluated in this randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients who undergo orthopedic surgery with duration of longer than one hour
* Patients with a history of ischemic heart disease (stable or unstable angina, myocardial infarction)
* American Society of Anesthesiology (ASA) Physical Status Classification of 1, 2, or 3

Exclusion Criteria:

* Peripheral vascular disease involving upper or lower extremity
* Orthopedic surgery which uses the tourniquet

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Troponin-I | postoperative day one

SECONDARY OUTCOMES:
Cardiac enzyme blood level (Creatinine Kinase, Creatinine Kinase -Myocardial Band) | immediate postoperative
Cardiac enzyme blood level (Creatinine Kinase, Creatinine Kinase -Myocardial Band) | postoperative day one
Cardiac enzyme blood level (Creatinine Kinase, Creatinine Kinase -Myocardial Band) | postoperative day two
Cardiac enzyme blood level (Creatinine Kinase, Creatinine Kinase -Myocardial Band) | postoperative day four
Acute kidney injury | postoperative 48 hours
  Acute kidney injury determined by AKIN criteria
ST-II segment analysis by Electrocardiography | every 30 minutes during surgery
Oxygenation index (PaO2/FiO2) | 5 minutes after anesthesia induction
Oxygenation index (PaO2/FiO2) | 5 minutes before the end of surgery
Oxygenation index (PaO2/FiO2) | 20 minutes after the end of surgery
  (at PACU)
Oxygenation index (PaO2/FiO2) | postoperative day one
length of hospital stay | up to 24 week
  length of hospital stay
length of ICU stay | up to 24 week
  length of ICU stay
Postoperative wound infection | up to 24 week
  Postoperative wound infection
Postoperative incidence of pneumonia | up to 24 week
  Postoperative incidence of pneumonia
Postoperative incidence of myocardial ischemic event | up to 24 week
  Postoperative incidence of myocardial ischemic event
Troponin-I | immediate postoperative
Troponin-I | Postoperative day two
Troponin-I | Postoperative day four
Creatinine | Immediate Postoperative
Creatinine | Postoperative day one
Creatinine | Postoperative day two
Creatinine | Postoperative day four

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No